CLINICAL TRIAL: NCT01881425
Title: A Randomized Study Comparing the Safety and Efficacy of the InnFocus MicroShunt® Glaucoma Drainage System to Standard Trabeculectomy In Subjects With Primary Open Angle Glaucoma
Brief Title: InnFocus MicroShunt Versus Trabeculectomy Study
Acronym: IMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnFocus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INN005
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Primary Open Angle Glaucoma
Keywords: POAG
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- InnFocus MicroShunt (Experimental): InnFocus MicroShunt
  Interventions: Device: InnFocus MicroShunt
- Trabeculectomy (Active Comparator): glaucoma surgery to reduce IOP
  Interventions: Procedure: Glaucoma Surgery

INTERVENTIONS:
Procedure: Glaucoma Surgery — An initial pocket is created under the conjunctiva and Tenon's capsule and the wound bed is treated for two minutes with mitomycin C (MMC, 0.2 mg/ml)soaked sponges. This is done using a "fornix-based" conjunctival incision at the corneoscleral junction. A partial thickness scleral flap with its base at the corneoscleral junction after cauterization of the flap area, and a window opening is created under the flap with a Kelly-punch to remove a portion of the sclera, Schlemm's canal and the trabecular meshwork to enter the anterior chamber. An iridectomy is done in many cases to prevent future blockage of the sclerostomy. The scleral flap is then sutured loosely back in place with several sutures. The conjunctiva is closed in a watertight fashion at the end of the procedure.
  Arms: Trabeculectomy
Device: InnFocus MicroShunt — An initial pocket is created under the conjunctiva and Tenon's capsule and the wound bed is treated for two minutes with mitomycin C (MMC, 0.2 mg/ml)soaked sponges. This is done using a "fornix-based" conjunctival incision at the corneoscleral junction. After cauterization of the flap area, a knife is used to create a shallow pocket at the scleral surface and an opening into the AC. The device is then threaded through the track until the proximal end is in the anterior chamber and the fin of the device is pushed into the shallow scleral pocket. The device is checked to observe aqueous flow and the distal end placed under the Tenons/conjunctiva. The conjunctiva is closed in a watertight fashion at the end of the procedure.
  Arms: InnFocus MicroShunt

SUMMARY:
Assess the safety and effectiveness of the InnFocus MicroShunt when used to lower intraocular pressure (IOP) in subjects with primary open angle glaucoma where the IOP is not controlled when using maximum tolerated glaucoma medications.

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomized, controlled, multicenter, study. After informed consent is obtained, patients will be evaluated for eligibility based on glaucoma severity, eye health, and visual acuity.

Clinical follow up will be scheduled over the course of the 24 month study, and examinations will be repeated to monitor eye health. At the 1 and 2 year follow up, diurnal (IOP taken in the morning, mid-day, and afternoon in the same day) IOP evaluation will be done. Annual follow up will occur up to 2 years. The primary effectiveness endpoint is 20% or greater reduction in IOP from pre-op medicated IOP at 12 months.

ELIGIBILITY:
Inclusion Criteria: - POAG on maximum tolerated glaucoma meds - Medicated ≥15mmHg and ≤40mmHg - Exclusion Criteria: - Previous conjunctival incisional ophthalmic surgery - Anticipated need for additional ocular surgery during the study - Secondary glaucoma - Any condition that prevents the device implantation or trabeculectomy in the superior region of the study eye

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Palmberg, M.D., Ph.D., Study Director — Bascom Palmer Eye Institute
Locations (29):
- United States (24):
  - Eye Physicians and Surgeons of Arizona, Glendale, Arizona
  - Arizona Eye Consultants, Tucson, Arizona
  - Vold Vision, Fayetteville, Arkansas
  - University of California at Davis Eye Center, Davis, California
  - UCLA Jules Stein Eye Institute, Los Angeles, California
  - Ophthalmic Consultants of Connecticut, Fairfield, Connecticut
  - Inter-Mountain Eye Care, Eagle, Idaho
  - Chicago Glaucoma Consultants and CGC Eye Center, Glenview, Illinois
  - Eugene and Marilyn Glick Eye Institute, Indianapolis, Indiana
  - Stiles Eyecare Excellence, Overland Park, Kansas
  - Washington Eye Physicians and Surgeons, Chevy Chase, Maryland
  - Minnesota Eye Consultants, PA, Bloomington, Minnesota
  - Midwest Eye Surgery Center, Omaha, Nebraska
  - New York Eye and Ear Infirmary of Mt. Sinai, New York, New York
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Ophthalmic Surgeons and Consultants of Ohio, Columbus, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Ophthalmic Partners of Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Glaucoma Associates of Texas, Dallas, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - The Robert Cizik Eye Clinic, Houston, Texas
  - Rashid, Rice, Flynn and Reilley Eye Associates, San Antonio, Texas
  - Specialty Eye Care, Bellevue, Washington
- Pole Ophtalmologique de la Clinique Mutualiste, Pessac, Bordeaux, France
- Pisa University Hospital Cisanello, Pisa, Italy
- University Eye Clinic Maastricht, Maastricht, Netherlands
- Hospital Clínico San Carlos, Madrid, Spain
- Moorfields Eye Hospital, London, United Kingdom

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740
- [Derived] Baker ND, Barnebey HS, Moster MR, Stiles MC, Vold SD, Khatana AK, Flowers BE, Grover DS, Strouthidis NG, Panarelli JF; INN005 Study Group. Ab-Externo MicroShunt versus Trabeculectomy in Primary Open-Angle Glaucoma: One-Year Results from a 2-Year Randomized, Multicenter Study. Ophthalmology. 2021 Dec;128(12):1710-1721. doi: 10.1016/j.ophtha.2021.05.023. Epub 2021 May 27. PMID 34051211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents data for 527 out of 732 patients who were enrolled in the INN-005 study and who were either randomized to the MicroShunt or Trabeculectomy.
Groups:
- InnFocus MicroShunt: The treatment group consists of subjects who receive the InnFocus MicroShunt with Mitomycin C (MMC).
- Trabeculectomy: The control group consists of subjects who receive trabeculectomy with MMC
Period: Overall Study
Arm/Group | InnFocus MicroShunt | Trabeculectomy
Started | 395 | 132
Completed | 370 | 123
Not Completed | 25 | 9
Not completed — Death | 5 | 1
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Adverse Event | 3 | 0
Not completed — General Anesthesia panic attack | 0 | 1
Not completed — Subject randomized after study treatment cut off | 0 | 1
Not completed — Lost to Follow-up | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | InnFocus MicroShunt | Trabeculectomy | Total
Number analyzed (Participants) | 395 | 132 | 527
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 164 | 51 | 215
  >=65 years | 231 | 81 | 312
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 59 | 273
  Male | 181 | 73 | 254
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 11 | 82
  White | 311 | 113 | 424
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 13 | 5 | 18
  United States | 337 | 113 | 450
  Italy | 10 | 3 | 13
  United Kingdom | 10 | 5 | 15
  France | 12 | 2 | 14
  Spain | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With > 20% Decrease in Mean Diurnal Intraocular Pressure
Description: The primary effectiveness outcome is ≥ 20% reduction in mean diurnal IOP without increasing number of glaucoma medications from baseline to 12 months follow-up
Time Frame: 12 months
Population: Primary Effectiveness Endpoint at 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | InnFocus MicroShunt | Trabeculectomy
Number analyzed (Participants) | 395 | 132
Participants | 216 | 96

2. Primary Outcome: Number of Participants With > 20% Decrease in Diurnal Intraocular Pressure
Description: The primary effectiveness outcome is ≥ 20% reduction in mean diurnal IOP without increasing number of glaucoma medications from baseline to 24 months follow-up
Time Frame: 24 months
Population: Primary Effectiveness Endpoint at 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | InnFocus MicroShunt | Trabeculectomy
Number analyzed (Participants) | 395 | 132
Participants | 200 | 85

3. Secondary Outcome: Mean Diurnal Intraocular Pressure Change
Description: Secondary Effectiveness Endpoint #1 is the mean diurnal change in IOP from Screening at 12 months.
Time Frame: 12 months
Population: Intent-to-treat (ITT) Population consisted of 527 randomized subjects and was population for Primary Effectiveness Endpoint/Secondary Effectiveness Endpoint #2. 395 in MicroShunt group and 132 in Trab. Secondary Effectiveness Endpoint #1 based on Glaucoma Reoperation Censored Subpopulation ITT Population which is why numbers differ. Glaucoma Reoperation Censored Subpopulation (subject data excluded from date of a qualifying glaucoma reoperation).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | InnFocus MicroShunt | Trabeculectomy
Number analyzed (Participants) | 332 | 114
mmHg | -6.46 (5.56) | -9.80 (5.92)

4. Secondary Outcome: Mean Diurnal Intraocular Pressure Change
Description: Secondary Effectiveness Endpoint #1 is the mean diurnal change in IOP from Screening at 24 months
Time Frame: 24 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | InnFocus MicroShunt | Trabeculectomy
Number analyzed (Participants) | 301 | 110
mmHg | -6.55 (5.47) | -9.85 (5.48)

5. Secondary Outcome: Number of Participants With Postoperative Interventions at 12 Months
Description: The Secondary Effectiveness Endpoint #2 was having any physical or medical postoperative intervention (other than eye massage) intended to alter IOP by the Month 12 follow-up visit.
Time Frame: 12 months
Population: To show Postoperative Interventions at 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | InnFocus MicroShunt | Trabeculectomy
Number analyzed (Participants) | 395 | 132
Participants | 161 | 89

6. Secondary Outcome: Participants With Postoperative Interventions at 24 Months
Description: The Secondary Effectiveness Endpoint #2 was having any physical or medical postoperative intervention (other than eye massage) intended to alter IOP by the Month 24 follow-up visit.
Time Frame: 24 months
Population: To show Postoperative Interventions at 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | InnFocus MicroShunt | Trabeculectomy
Number analyzed (Participants) | 395 | 132
Participants | 219 | 93

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious Adverse Events (SAEs) were reported for the duration of the study (24 Months). This analysis population includes all subjects who were treated.
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device.
Arm/Group | InnFocus MicroShunt | Trabeculectomy
All-Cause Mortality (participants affected / at risk) | 5/395 | 1/131
Serious Adverse Events (participants affected / at risk) | 13/395 | 3/131
Other Adverse Events (participants affected / at risk) | 366/395 | 122/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | InnFocus MicroShunt (N=395) | Trabeculectomy (N=131)
Increased IOP Requiring Treatment (Eye disorders) | 7 | 0
Retinal Complication (Dialysis, Flap Tears, Detachment, Decompression or Proliferative Retinopathy) (Eye disorders) | 1 | 2
Aqueous Humor Misdirection (malignant glaucoma) (Eye disorders) | 1 | 0
Choroidal Effusion / Detachment (Eye disorders) | 1 | 0
Hypotony (IOP < 6mmHg at any Time) (Eye disorders) | 1 | 0
Loss 2 or More Lines of BCVA on 2 Consecutive Standard Follow-ups 90 Days or more after Implantation (Eye disorders) | 1 | 0
Subconjunctival Bleeding or Hyphema at any time (including Microhyphema) (Eye disorders) | 0 | 1
Glaucoma Progression with Vision Loss (Eye disorders) | 1 | 0
Confirmed Worsening in the Visual Field (Eye disorders) | 1 | 0 — Confirmed Worsening in the Visual Field Mean Deviation (MD) of ≥ 2.5 DB compared to MD used to determine Subject Eligibility (confirmed on at least 2 out of 3 Visual Field Tests performed after 3 Months Post Procedure)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | InnFocus MicroShunt (N=395) | Trabeculectomy (N=131)
Increased IOP Requiring Treatment (Eye disorders) | 215 | 73
Hypotony (IOP < 6mmHg at any Time) (Eye disorders) | 121 | 67
Subconjunctival Bleeding or Hyphema at any time including Microhyphema (Eye disorders) | 83 | 23
Confirmed Worsening in the Visual Field Mean Deviation (Eye disorders) | 73 | 27 — Confirmed Worsening in the Visual Field Mean Deviation (MD) of ≥ 2.5 DB compared to MD used to determine Subject Eligibility (confirmed on at least 2 out of 3 Visual Field Tests performed after 3 Months Post Procedure)
Cataract Progression (Eye disorders) | 56 | 28
Loss 2 or More Lines of BCVA (Eye disorders) | 55 | 23 — Loss 2 or More Lines of BCVA on 2 Consecutive Standard Follow-ups 90 Days or more after Implantation (excluding Posterior Capsule Opacification, followed by post Nd: YAG Capsulotomy and improvement in BCVA)
Bleb Leak / Bleb Leak Based on Positive Seidel Test (Eye disorders) | 36 | 19
Corneal Edema (Eye disorders) | 35 | 8
Anterior Chamber Cells and/or Flare (Eye disorders) | 31 | 11
Dry Eye (Eye disorders) | 28 | 12
Pain (Eye disorders) | 26 | 13
Blurry Vision (Eye disorders) | 33 | 9
Shallow Anterior Chamber (Eye disorders) | 27 | 11
Foreign Body Sensation (Eye disorders) | 30 | 10
Ptosis (Eye disorders) | 33 | 7
Bleb Related Complications (Eye disorders) | 28 | 9
Choroidal Effusion / Detachment (Eye disorders) | 18 | 10
Diplopia (Eye disorders) | 26 | 7
Conjunctival Injection / Conjunctival Hyperemia / Conjunctival Inflammation / Conjunctival Scarring (Eye disorders) | 23 | 6
Encapsulated Bleb (Eye disorders) | 23 | 3
Ocular Irritation (Eye disorders) | 18 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT01881425/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT01881425/SAP_001.pdf